CLINICAL TRIAL: NCT05696626
Title: An Open Label, Randomized, Multicenter Study Comparing the Efficacy and Safety of the Combination of Lasofoxifene and Abemaciclib to the Combination of Fulvestrant and Abemaciclib for the Treatment of Pre- and Postmenopausal Women and Men With Locally Advanced or Metastatic ER+/HER2- Breast Cancer With an ESR1 Mutation
Brief Title: Evaluation of Lasofoxifene Combined With Abemaciclib Compared With Fulvestrant Combined With Abemaciclib in Locally Advanced or Metastatic ER+/HER2- Breast Cancer With an ESR1 Mutation
Acronym: ELAINEIII
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sermonix Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMX 22-002
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lasofoxifene; abemaciclib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: open label, randomized, parallel-group, multicenter study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Pre- and Postmenopausal Women and Men with locally advanced or metastatic ER+/HER2- breast cancer who have disease progression on an AI in combination with either palbociclib or ribociclib as their first hormonal treatment for metastatic disease and who have an ESR1 mutation.
  Interventions: Drug: Lasofoxifene in combination with abemaciclib
- Reference Therapy (Active Comparator): Pre- and Postmenopausal Women and Men with locally advanced or metastatic ER+/HER2- breast cancer who have disease progression on an AI in combination with either palbociclib or ribociclib as their first hormonal treatment for metastatic disease and who have an ESR1 mutation.
  Interventions: Drug: Fulvestrant in combination with abemaciclib

INTERVENTIONS:
Drug: Lasofoxifene in combination with abemaciclib — 5 mg/d of oral lasofoxifene plus oral abemaciclib 150 mg twice a day
  Arms: Treatment
Drug: Fulvestrant in combination with abemaciclib — Fulvestrant 500 mg intramuscular (IM) on Days 1, 15, and 29 and then once monthly thereafter plus oral abemaciclib 150 mg twice a day
  Arms: Reference Therapy

SUMMARY:
The goal of this clinical trial is to assess the efficacy, safety and tolerability of the combination of lasofoxifene and abemaciclib compared to fulvestrant and abemaciclib for the treatment of pre- and postmenopausal women and men who have previously received ribociclib or palbociclib-based treatment and have locally advanced or metastatic estrogen receptor positive (ER+)/human epidermal growth factor 2 negative (HER2-) breast cancer with an estrogen receptor 1 (ESR1) mutation.

The main question the study aims to answer is:

• To compare the efficacy of the combination of lasofoxifene and abemaciclib with that of fulvestrant and abemaciclib Participants will receive either receive 5 mg/d of oral lasofoxifene plus oral abemaciclib 150 mg twice a day or the combination of fulvestrant 500 mg intramuscular (IM) on Days 1, 15, and 29 and then once monthly thereafter plus oral abemaciclib 150 mg twice a day.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- or postmenopausal women or men.
2. Locally advanced and/or metastatic ER+ breast cancer with radiological or clinical evidence of progression on an AI in combination with either palbociclib or ribociclib as their first hormonal treatment for metastatic disease.
3. Histological or cytological confirmation of ER+/HER2 - disease
4. No evidence of progression for at least 6 months on an AI/CDKi combination for advanced breast cancer.
5. At least 1 or more ESR1 point mutations in the ESR1 ligand binding domain as assessed in cell- free ctDNA obtained from a blood or breast cancer tissue.
6. Locally advanced or metastatic breast cancer with either measurable (according to RECIST 1.1) or non-measurable lesions.
7. Subjects may have received 1 cytotoxic chemotherapy regimen in the metastatic disease setting prior to study entry, but must have recovered from chemotherapy acute toxicity excluding alopecia and Grade 2 peripheral neuropathy.
8. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
9. Adequate organ function
10. Able to swallow tablets
11. Brain metastases are allowed only if the following 4 parameters hold:

    1. Asymptomatic,
    2. Definitively treated (e.g., radiotherapy, surgery),
    3. Not requiring steroids up to 4 weeks before study treatment initiation, AND
    4. Central nervous system disease stable for >3 months prior to registration as documented by magnetic resonance imagining (MRI).
12. Able to understand and voluntarily sign a written informed consent before any screening procedures.
13. Every attempt should be made to obtain a biopsy of metastatic breast cancer tissue, when safe and feasible, to provide histological or cytological confirmation of ER+/HER2- disease as assessed by a local laboratory, according to American Society of Clinical Oncology/College of American Pathologists guidelines, using slides, paraffin blocks, or paraffin samples. If a biopsy is done, it may undergo genomic testing at some point to assess for ESR1 mutations and correlation with ctDNA results. If a biopsy is not possible or inappropriate from a clinical standpoint, the ER and HER2 status from the subject's most recent biopsy must confirm that the subject is ER+ and HER2

Exclusion Criteria:

1. Lymphangitic carcinomatosis involving the lung.
2. History of Grade 3 or Grade 4 interstitial lung disease (ILD) on previous therapy.
3. Visceral crisis in need of cytotoxic chemotherapy as assessed by the investigator.
4. Prior progression of disease on abemaciclib, fulvestrant, or other selective estrogen receptor degrader (SERD) therapy.
5. Subjects with a known hypersensitivity to fulvestrant or to any of the excipients
6. Radiotherapy within 30 days prior to Visit 0 (Day 1) except in case of localized radiotherapy for analgesic purposes or for lytic lesions at risk of fracture, which can then be completed within 7 days prior to Visit 0 (Day 1). Subjects must have recovered from radiotherapy toxicities prior to Visit 0 (Day 1).
7. Known RB1 mutations or deletions that in the opinion of the investigator confer resistance to CDK4/6i. (Screening for RB1 mutation is not required for entry.)
8. History of long QTc (Q-T interval corrected for heart rate) syndrome or a QTc of >480 msec.
9. History of a pulmonary embolus (PE), deep vein thrombosis (DVT), or any known thrombophilia, unless the event occurred greater than 6 months prior to screening and the subject is treated with chronic anticoagulant therapy such as apixaban (Eliquis) or rivaroxaban (Xarelto).
10. Lasofoxifene is not recommended for use in subjects with conditions that place them at increased risk for VTEs (such as severe congestive heart failure [CHF] or prolonged immobilization).
11. On concomitant strong CYP3A4 inhibitors.
12. On strong and moderate CYP3A4 inducers.
13. Any significant co-morbidity that would impact the study or the subject's safety, including subjects with significant malabsorption.
14. Active systemic bacterial or fungal infection (requiring intravenous [IV] antibiotics or antifungals at the time of initiating study treatment).
15. Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
16. History of malignancy within the past 5 years (excluding breast cancer), except basal cell or squamous cell carcinoma of the skin curatively treated by surgery.
17. Positive serum pregnancy test (only if premenopausal).
18. Sexually active premenopausal women and men unwilling to use double-barrier contraception.
19. Women who are breast feeding
20. History of non-compliance to medical regimens.
21. Unwilling or unable to comply with the protocol.
22. Current participation in any clinical research trial involving an investigational drug or device within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Within approximately 3 years
  PFS is defined as the time from the date of randomization [Visit 0 (Day 1)] to the earliest date of first documented progression per RECIST 1.1 or death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Within approximately 3 years
  ORR is defined as the percentage of subjects with measurable disease at baseline whose best overall response is either a confirmed CR or a confirmed PR according to RECIST 1.1.
Overall survival (OS) | Within approximately 3 years
  Overall survival is defined as time from the date of Visit 0 (Day 1) to death due to any cause.
Clinical benefit rate (CBR) | Within approximately 3 years
  CBR is defined as the percentage of subjects with best overall response of confirmed CR, confirmed PR, or stable disease (SD) with a duration of 24 weeks or longer according to RECIST 1.1. As used in this calculation, stable disease is defined as stable disease in those subjects with measurable disease plus nonPR/non progressive disease (PD) in subjects with non-measurable disease.
Duration of response (DoR) in subjects with an objective response | Within approximately 3 years
  DoR is from the date of first documented confirmed response (CR or PR) to the date of first documented progression of disease or death due to any cause, whichever is earlier.
Time to response (TTR) in subjects with an objective response | Within approximately 3 years
  TTR is from the date of randomization to the date of first documented confirmed response (CR or PR).
Time to cytotoxic chemotherapy | Within approximately 3 years
  From the date of randomization to the date of first documented use of cytotoxic chemotherapy.
Quality of Life (QoL) evaluated using the Functional Assessment of Cancer Therapy-Breast Cancer-Endocrine Subscale (FACT B-ES) | Within approximately 3 years
  Scale ranges from 'Not at all' to 'Very much'
Incidence of Adverse Events (AEs) and Serious AEs | Within approximately 3 years
  The type, severity (graded by Common Terminology Criteria for Adverse Events [CTCAE version 5.0]), course, duration, seriousness, and relationship to study treatment will be assessed at each visit

CONTACTS AND LOCATIONS:
Locations (222):
- United States (35):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - University of Arizona - Cancer Center, Tucson, Arizona
  - Providence Medical Foundation - Santa Rosa, CA, Santa Rosa, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Miami Cancer Institute Plantation, Plantation, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Allina Health System DBA Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Renown Regional Medical Centre, Reno, Nevada
  - Cancer Care Specialists, Reno, Nevada
  - New Jersey Cancer Care, PA, Belleville, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Presbyterian Rust Cancer Center, Rio Rancho, New Mexico
  - The Blavatnik Family - Chelsea Medical Center at Mount Sinai, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Altru Health Systems, Grand Forks, North Dakota
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center - Arthur G. James Cancer Hospital and Richard J. Solovev Research Institute (OSUCCC - James), Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas
  - Swedish Cancer Institute (SCI), Seattle, Washington
- Australia (3):
  - Blacktown Hospital, Blacktown
  - Concord Repatriation General Hospital, Concord
  - Mater Misericordiae Ltd, South Brisbane, South Brisbane
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital (UZA), Edegem
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHU UCL Namur - Site De Sainte-Elisabeth, Namur
- Canada (5):
  - The Ottawa General Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre -Bayview Campus, Toronto, Ontario
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Lady Davis Institute for Medical Research Jewish General Hospital, Montreal, Quebec
  - CIUSSS du Saguenay-Lac-Saint-Jean, Saguenay, Quebec
- China (77):
  - Anhui Provincial Cancer Hospital, Anhui
  - Anyang Tumour Hospital, Anyang
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqicun
  - The Second Hospital of Dalian Medical University, Dalian
  - Deyang People's Hospital, Deyang
  - Fuyang Cancer Hosptial, Fuyang
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Zhujiang Hospital of Nanfang Medical University, Guandong
  - Guangdong Provincial People's Hospital, Guangdong
  - Meizhou People's Hospital, Guangdong
  - Peking University Shenzhen Hospital, Guangdong
  - Sun Yat-Sen University- Cancer Center, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou
  - Hebei Medical University - The Fourth Hospital - Hebei Provincial Tumor Hospital, Hebei
  - Xiangyang Central Hospital, Hubei
  - Xiangya Hospital Central South University, Hunan
  - Jieyang People's Hospital, Jieyang
  - Shandong Province Tumor Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Gansu Provincial Hospital, Lanzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - Linyi Cancer Hospital, Linyi
  - Luoyang Central Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The Affiliated Hospital of Southwest Medical University (Luzhou Medical College), Luzhou
  - Jiangxi Cancer Hospital, Nanchang
  - Nanchang People's Hospital, Nanchang
  - Jiangsu Province Hospital - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Nanyang Central Hospital, Nanyang
  - The Second People's Hospital of Neijiang, Neijiang
  - Ningbo Medical Center Li Huili Hospital, Ningbo
  - The First People'S Hospital of Ping Ding Shan, Pingdingshan
  - Qingdao Central Hospital, University of Health and Rehabilitation Sciences, Qingdao
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Quanzhou First Hospital, Quanzhou
  - Huashan Hospital, Fudan University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Cancer Center, Shang’ai
  - First Affiliated Hospital of Xi'an Jiaotong University, Shanxi
  - The Central Hospital of Shaoyang, Shaoyang
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Yuebei People's Hospital, Shouguang
  - University of Electonic Science & Technology (UESTC) - Sichuan Cancer Hospital & Institute, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technolog, Wuhan
  - The Second People's Hospital of WuHu, Wuhu
  - The First Affiliated Hospital of Air Force Medical University, Xi Ail
  - The first affiliated hospital of Xiamen University, Xiamen
  - Zhongshang Hospital Xiamen University, Xiamen
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xinzheng
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Yuncheng Central Hospital, Yuncheng
  - Zhejiang cancer hospital, Zhejiang
  - Zhejiang Provincial People's Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhongshan City People's Hospital, Zhongshan
  - Zhumadian Central Hospital, Zhumadian
- France (13):
  - Institut Sainte Catherine, Avignon
  - Service d'Oncologie Medicale - CHRU Besancon, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Groupement de Cooperation Sanitaire (GCS) ELSAN - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers - Pole Regional de Cancerologie de Poitiers (PRC), Poitiers
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Klinikum rechts der Isar der Technischen Universitaet Muenchen, München
- Israel (10):
  - Haemek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Ein-Karem Medical Center, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (14):
  - Azienda Ospedaliero-Universitaria delle Marche, Ancona
  - Centro Riferimento Oncologico - Aviano, Aviano
  - La Fondazione e l'Istituto di Candiolo, Candiolo
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori - IRST S.r.l., Meldola
  - Istituto Europeo di Oncologia, Milan
  - Humanitas Istituto Clinico Catanese, Misterbianco
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero Universitaria Maggiore Della Carita, Novara
  - Istituto Oncologico Veneto-I.R.C.C.S. - Ospedale Busonera, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale Borgo Trento, Verona
- Poland (8):
  - KO - MED Centra Kliniczne Sp. z o.o., Wojewodzki Szpital Specjalistyczny w Bialej Podlaskiej, Biała Podlaska
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Oddzial w Gliwicach, I Klinika Radioterapii i Chemioterapii, Gliwice
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Oddzial Onkologii Klinicznej, Krakow
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie - Oddzial Onkologii Klinicznej z Pododdzialem Dziennym, Krakow
  - Instytut Centrum Zdrowia Matki Polki - Klinika Onkologii, Lodz
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Oddzial Chemioterapii, Poznan
  - Wielkopolskie Centrum Onkologii (WCO) / The Greater Poland Cancer Center, Poznan
  - Mazowiecki Szpital Onkologiczny, Wieliszew
- Romania (6):
  - Centrul Medical Focus, Bucharest
  - Radiotherapy Center Cluj, Cluj-Napoca
  - Onco Clinic Consult SA, Craiova
  - Oncology Center Sfantul Nectarie, Craiova
  - Gral Medical SRL, Piteşti
  - OncoMed Oncology Center, Timișoara
- Curie Oncology, Singapore, Singapore
- South Korea (5):
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (13):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Beata Maria Ana, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (7):
  - Changhua Christian Hospital (CCH), Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Taoyuan
- Turkey (Türkiye) (10):
  - Liv Hospital Ankara, Çankaya, Ankara
  - Istanbul University CAPA Medical Faculty, Çapa, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Kadiköy, Istanbul
  - Ege University Medical Faculty Hospital, Bornova, İzmir
  - Suat Seren Training and Research Hospital, Konak, İzmir
  - Kocaeli University Research and Application Hospital, İzmit, Kocaeli
  - Ankara University Medical Faculty Medical Oncology Department, Ankara
  - Uludag University Faculty of Medicine Hospital, Bursa
  - Trakya University Medical Faculty Hospital, Edirne
  - Medical Point Izmir Hospital, Izmir
- United Kingdom (9):
  - Velindre Cancer Center, Cardiff
  - Princess Alexandra Hospital - Harlow, Harlow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Free London NHS Foundation Trust, London
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Milton Keynes Hospital, Milton Keynes
  - Nottingham City Hospital, Nottingham
  - University Hospital of North Tees, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goetz MP, Wander SA, Bachelot T, de Nonneville A, Gal-Yam EN, Sammons SL, Shen S, Twelves C, Boruta G, Portman DJ, Damodaran S. ELAINE 3: phase 3 study of lasofoxifene plus abemaciclib to treat ER+/HER2-, ESR1-mutated, metastatic breast cancer. Future Oncol. 2025 May;21(11):1317-1324. doi: 10.1080/14796694.2025.2481825. Epub 2025 Apr 13. PMID 40222048